CLINICAL TRIAL: NCT03888482
Title: Clinical Comparison of DDT2 Contact Lens and a Daily Disposable Contact Lens - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLE383-C010
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Refractive Error; Myopia
Keywords: Visual acuity; VA; Daily disposable contact lenses
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- DDT2, then Clariti (Other): Verofilcon A contact lenses worn first, with somofilcon A contact lenses worn second, as randomized. Each product was worn bilaterally (in both eyes) for 8 -1/+2 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Somofilcon A contact lenses
- Clariti, then DDT2 (Other): Somofilcon A contact lenses worn first, with verofilcon A contact lenses worn second, as randomized. Each product was worn bilaterally (in both eyes) for 8 -1/+2 days in a daily disposable modality.
  Interventions: Device: Verofilcon A contact lenses; Device: Somofilcon A contact lenses

INTERVENTIONS:
Device: Verofilcon A contact lenses — Investigational daily disposable soft contact lenses
  Other Names: DDT2
Device: Somofilcon A contact lenses — Commercially available daily disposable soft contact lenses
  Other Names: clariti® 1 day; Clariti

SUMMARY:
The purpose of this study was to evaluate visual acuity at distance when wearing DDT2 contact lenses compared to Clariti contact lenses.

DETAILED DESCRIPTION:
Subjects were expected to attend 3 study visits and wear the DDT2 and Clariti study lenses in a crossover design for approximately 14 - 20 days (7 - 10 days for each product).

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Informed Consent Form that has been approved by an Institutional Review Board.
* Willing and able to attend all scheduled study visits as required per protocol.
* Current wearer of spherical soft contact lenses.

Key Exclusion Criteria:

* Any ocular condition that contraindicates contact lens wear.
* Previous or current habitual wearer of clariti® or DAILIES TOTAL1® contact lenses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CDMA Project Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Alcon Investigative Site, Jacksonville, Florida
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Orlando, Florida
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Powell, Ohio
  - Alcon Investigative Site, Warwick, Rhode Island
  - Alcon Investigative Site, Brentwood, Tennessee
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was performed at 8 study centers in the United States (US).
Pre-assignment Details: Of the 154 enrolled, 2 were exited from the study as screen failures and 1 subject was randomized but not exposed. This reporting group includes all exposed subjects (151).
Period: First Wear Period (8 -1/+2 Days)
Arm/Group | DDT2, Then Clariti | Clariti, Then DDT2
Started | 76 | 75
Completed | 76 | 75
Not Completed | 0 | 0
Period: Second Wear (8 -1/+2 Days)
Arm/Group | DDT2, Then Clariti | Clariti, Then DDT2
Started | 74 (2 subjects were discontinued between Treatment 1 and Treatment 2.) | 75
Completed | 73 | 74
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DDT2, Then Clariti | Clariti, Then DDT2 | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (7.9) | 31.8 (7.9) | 33.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 47 | 103
  Male | 20 | 28 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 73 | 69 | 142
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 65 | 67 | 132
  Black or African American | 5 | 1 | 6
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 1 | 2 | 3
  Multi-racial | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 76 | 75 | 151

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance Visual Acuity With Study Lenses
Description: Visual acuity was assessed and collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 8, each product
Population: Full analysis set (FAS): All randomized subjects/eyes with non-missing responses, who were exposed to any study lenses evaluated in this study, with the exception of the lenses used at Visit 1 for optimization and fitting.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- DDT2: Verofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
- Clariti: Somofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
Arm/Group | DDT2 | Clariti
Number analyzed (Participants) | 151 | 149
Number analyzed (eyes) | 294 | 296
logMAR | -0.08 (0.006) | -0.08 (0.006)
Statistical Analysis 1: Comparison: DDT2 vs Clariti; Test type: Non-Inferiority — Non-inferiority margin = 0.05; Mixed effects repeated measures model; Mixed effects repeated measures model with terms for lens, period and sequence as fixed effects and subject as a random effect; Least Squares Mean Difference = 0.00, 95% CI 1-sided [upper limit 0.01] — Difference = DDT2 - Clariti

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent to study exit (approximately 14-20 days). The safety analysis set included all subjects/eyes exposed to any study lenses evaluated in this study, with the exception of the lenses used at Visit 1 for the purpose of parameter optimization and fitting, as they were not intended for the assessment of safety.
Description: Adverse events (AEs) were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population of ocular AEs is reported in units of eyes; all other populations are reported in units of subjects.
Groups:
- DDT2 - Ocular; DDT2 - Systemic / Nonocular: Verofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
- Clariti - Ocular; Clariti - Systemic / Nonocular: Somofilcon A contact lenses worn bilaterally (in both eyes) during Period 1 or Period 2, as randomized, for 8 -1/+2 days in a daily disposable modality.
Arm/Group | DDT2 - Ocular | DDT2 - Systemic / Nonocular | Clariti - Ocular | Clariti - Systemic / Nonocular
All-Cause Mortality (participants affected / at risk) | 0/302 | 0/151 | 0/298 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/302 | 0/151 | 0/298 | 0/149
Other Adverse Events (participants affected / at risk) | 0/302 | 0/151 | 0/298 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2019-03-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03888482/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT03888482/SAP_001.pdf